CLINICAL TRIAL: NCT01438437
Title: Trial of Ablation of Small Hepatocellular Carcinomas in Patients of Cirrhosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Subrat Kumar Acharya, Proffessor and Head, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-16/11/2001
Record Dates: First submitted 2011-09-14; First posted 2011-09-22 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Radiofrequency ablation; Percutaneous acetic acid ablation; Tumour response
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneous acetic acid (Active Comparator)
  Interventions: Procedure: PAI
- Radiofrequency ablation (Active Comparator)
  Interventions: Procedure: RFA

INTERVENTIONS:
Procedure: PAI — Under local anaesthesia, taking proper aseptic precautions, 40% acetic acid (total dose not exceeding 3 times the diameter of the mass, (not more than 2ml in one sitting), will be injected into the mass through the percutaneous route
  Arms: Percutaneous acetic acid
Procedure: RFA — Under aseptic conditions and local anesthesia, the needle electrode would be introduced percutaneously into the tumor under ultrasound guidance.
  Arms: Radiofrequency ablation

SUMMARY:
The purpose of this study is to assess the efficacy of Radiofrequency ablation (RFA) and percutaneous acetic acid ablation (PAI) in the management of small hepatocellular carcinoma (HCC) in patients of cirrhosis of liver.

DETAILED DESCRIPTION:
Setting The study would be conducted at the All India Institute of Medical Sciences, New Delhi, a tertiary care teaching hospital, in the departments of Gastroenetrology and Radiodiagnosis.

Sample size Taking RFA as a standard procedure with an estimated success rate of 95%, a sample size of minimum 27 for each arm is required to detect an equivalence difference of 10%, assuming that PAI has a success rate of 85%. This sample size is expected to provide a power of 80%.

Randomization

* Stratified randomization of Child A and B will be done.
* Randomization into A (Acetic acid) and B (Radiofrequency ablation) will be done.

Diagnostic criteria

* Cirrhosis of liver- Diagnosis will be founded on the basis of clinical, biochemical, imaging and endoscopy findings.

Hepatocellular carcinoma- when any one of the following is present

1. Two imaging modalities (dual phase CT (DPCT)/ contrast enhanced Magnetic Resonance Imaging (MRI)) showing arterialization of the hepatic mass
2. AFP more than 400ng/ml along with arterialisation on one imaging modality (DPCT/ contrast enhanced MRI)
3. Fine needle aspiration cytology (FNAC)

Definitions

1. Local recurrence : When the Triple phase CT shows-

   * An area of nodular enhancement that abuts or surrounds the ablation defect or protrudes into the low attenuating necrotic tissue (may sometimes be seen only on arterial phase of CT)
   * Recurrent soft tissue causing distortion of the otherwise smooth interphase with the adjoining liver parenchyma.
2. Fresh lesion- When a new lesion is seen in the liver at a site other than the primary site of the treated lesion with normal liver parenchyma intervening in between will be considered as a fresh lesion.
3. Residual disease or incomplete ablation When the follow up Triple phase CT shows-

   * Residual nodular enhancement that abuts or surrounds the low attenuating ablation defect or protrudes into the low attenuating necrotic tissue (may sometimes be seen only on arterial phase of CT)
   * Residual soft tissue causing distortion of the otherwise smooth interphase with the adjoining liver parenchyma.
   * Concenteric hyperemia around the low attenuating defect showing area of focal nodularity or asymmetric thickness.
4. End point of ablation When the Triple phase CT shows-

   * A homogenous, well defined, uniformly low attenuating defect larger than the pretreatment size.
   * No residual soft tissue seen within or at the periphery of the low attenuating defect
   * Concentric hyperemia around the low attenuating defect of uniform thickness with no focal nodularity.

Follow up

1. Clinical follow up

   * All patients would be followed up in the Liver clinic monthly unless their clinical condition warrants earlier follow up
   * Liver function tests/ complete blood count would also be done at each visit and Alfafetoprotein (AFP) every six months
   * Patient tolerance, child's status would be estimated.
2. Imaging follow up

   * At one month, a dual phase CT would be done to ascertain the local response to therapy and the need to repeat the procedure. After achieving the end point after ablation (PAI and RFA, the DPCT would be done at 3 and 6 monthly intervals.

Duration of follow up - Since more than 80% recurrence occurs in 2 years therefore the duration of follow up would be 2 years after ablation.

ELIGIBILITY:
Inclusion Criteria:

* Child's A or B cirrhosis with liver mass.
* Number of liver masses not more than 5 and the size of each <5cm in diameter.
* No extrahepatic disease.
* Absence of malignant portal vein thrombosis.
* Platelet count more than 70,000/mm3
* Prothrombin time more than 50%.
* Written consent of patient.

Exclusion Criteria:

* Childs'C cirrhosis with liver mass.
* Liver mass >5cm in diameter.
* Number of liver masses more than 3
* Peripherally located masses with no hepatic parenchyma around
* Liver mass not discernable on ultrasound.
* Extra hepatic disease like RP adenopathy, distant metastasis.
* Coagulation disorders.
* Unwilling patient

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2001-03; Primary Completion 2014-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Local tumor response | 2 years

SECONDARY OUTCOMES:
Survival rate | 2 years
Number of patients with complications | 2 years
  Number of patients developing any complications during and after procedure will be noted.
Change from baseline in Child status at 1 year | 2 years
  Child status is calculated from the following 5 parameters
  1. Bilirubin < 2: 1, 2-3: 2 and > 3 : 3 points
  2. Albumin: > 3.5: 1, 2.8-3.5 : 2 and <2.8: 3 points
  3. Prothrombin time( seconds over control): 1-3: 1, 4-6: 2 and > 6: 3
  4. Encephalopathy: None: 1, (grade 1 and 2): 2 and (grade 3 and 4): 3
  5. Ascites: Absent: 1, slight: 2 and moderate: 3
  Child A: score 5-6, Child B: 7-9 and Child C: 10 or more

CONTACTS AND LOCATIONS:
Locations (1):
- AIIMS, New Delhi, National Capital Territory of Delhi, India